CLINICAL TRIAL: NCT05843292
Title: Short-term Sintilimab in Combination With Taxane and Carboplatin for Neoadjuvant Therapy in Triple-negative Breast Cancer, an Open-labeled, Single Arm Trial
Brief Title: Short-term Sintilimab in Combination With Taxane and Carboplatin for Neoadjuvant Therapy in Triple-negative Breast Cancer
Acronym: NeoSTEP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Innovent Biologics, Inc. (Other); CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Director of Comprehensive Breast Health Center, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoSTEP
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Triple-negative Breast Cancer
Keywords: Short-term Sintilimab; Taxane; Carboplatin; Neoadjuvant Therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — taxane; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-term Sintilimab in Combination With Taxane and Carboplatin (Experimental): Prior to surgery: 2 cycles of sintilimab, in combination with 4 cycles of taxane and carboplatin
  Interventions: Drug: Taxane and Carboplatin; Drug: Short-term Sintilimab; Procedure: Surgery

INTERVENTIONS:
Drug: Taxane and Carboplatin — Nab-paclitaxel 100mg/m2+ Carboplatin AUC2 by intravenous (IV) infusion on day1, day8 and day15, every 4 weeks, for 4 cycles.
  or Docetaxel 75mg/m2+ Carboplatin AUC5 by intravenous (IV) infusion on day1, every 3 weeks, for 4 cycles.
  or Paclitaxel 80mg/m2+ Carboplatin AUC2 by intravenous (IV) infusion on day1, day8 and day15, every 4 weeks, for 4 cycles.
Drug: Short-term Sintilimab — Sintilimab 200mg by intravenous (IV) infusion on day1, every 3 weeks, for 2 cycles.
Procedure: Surgery — All participants who are eligible for surgery will undergo surgery and have their pathologic response evaluated.

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of short-term sintilimab in combination with taxane and carboplatin for neoadjuvant therapy in female early-stage triple-negative breast caner patients aging from 18 to 70 years with unilateral and invasive primary lesions above 1cm. The main questions it aims to answer are:

1. Does short-term sintilimab in combination with taxane and carboplatin lead to acceptible pathological complete response (pCR) rates, objective response rates (ORR), event-free survival (EFS) and overall survival (OS)?
2. Does short-term sintilimab in combination with taxane and carboplatin lead to less adverse events than regular-term ICIs reported in literature?

Participants will be given 2 cycles of sintilimab, in combination with 4 cycles of taxane and carboplatin before surgery. An optional core-needle biopsy is performed after completing 2 cycles of sintilimab. All participants will be given regular follow-up post surgery according to ASCO guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years, female;
2. Unilateral, invasive, primary breast cancer, T≥1cm, cN0-3, M0;
3. Immunohistochemistry(IHC): ER, PR<10%; HER-2 IHC "0", OR IHC "+", OR IHC "++" AND fluorescence in situ hybridization (FISH) negative;
4. At least one measurable lesion according to RECIST V1.1;
5. Newly or recently-collected core needle biopsy specimen of the primary lesion available for PD-L1 status determination;
6. ECOG score 0 or 1 within 10 days prior to drug administration;
7. Currently not pregnant or breastfeeding, and meet at least one of the following conditions:

   1. NOT women of childbearing potential (WOCBPs).
   2. WOCBPs that strictly adopt contraceptive measures during treatment and within at least 6 months after last drug administration.
8. Organs well-functioned according to laboratory examination and imaging;
9. Having good compliance with treatment plans, being capable of understanding the research process, and having signed a written informed consent.

Exclusion Criteria:

1. Bilateral invasive breast cancer or metastatic (Stage IV) breast cancer;
2. With severe cardiovascular conditions:

   1. Myocardial infarction, acute coronary syndrome or PCI/CABG within 6 months;
   2. Current NYHA II-IV congestive heart failure (CHF) or past history of NYHA III-IV CHF.
3. Immunodeficiency, or undergoing systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to drug administration;
4. Active autoimmune diseases requiring systemic treatment within the past 2 years;
5. Known history of active tuberculosis caused by Bacillus Tuberculosis;
6. History of non infectious pneumonia requiring steroid treatment, or active pneumonia of all types;
7. Severe systemic infections, or other serious illnesses;
8. History of other malignant tumors within the past 5 years, except cured cervical carcinoma in situ and non-melanoma skin cancer;
9. Known history of human immunodeficiency virus (HIV) infection;
10. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection;
11. Known allergy or intolerance to therapeutic drugs or their excipients;
12. History of receiving cytotoxic chemotherapy, endocrine therapy, biological therapy or radiation therapy for any reason;
13. History of receiving anti PD-1, anti PD-L1, or anti PD-L2 drugs; or targeted drugs that act on stimulating or co-inhibitory T cell receptors (CTLA-4, OX 40, CD137 etc.);
14. Enrolled in a study of an investigational drug/instrument and given intervention within 4 weeks prior to drug administration for regular drugs/instruments and within 12 months for anticancer or anti-proliferative drugs/instruments;
15. Live vaccine (including but not limited to the following: measles, mumps, rubella, chickenpox/shingles, yellow fever, rabies, BCG, typhoid vaccines, and nasal influenza vaccines such as FluMist®) inoculation within 30 days prior to drug administration;
16. History of mental illness or drug abuse that may affect compliance with trial requirements;
17. During pregnancy or breastfeeding, or WOCABs that refuse to adopt strict contraceptive measures;
18. Deemed to be not appropriate for participating in this study by researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rates | At surgery.
  The percentage of participants with the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes after completion of neoadjuvant therapy and surgery (that is, ypT0/is, ypN0, in accordance with the current American Joint Committee on Cancer [AJCC] staging system).

SECONDARY OUTCOMES:
Objective Response Rates (ORR) | At surgery.
  The percentage of participants with complete response (CR) and partial response (PR) in accordance with RECIST V1.1 definitions.
Event-free survival (EFS) | From Baseline to EFS event or date last known to be alive and event-free (up to 10 years)
  EFS is defined as the time from diagnosis to the first documentation of one of the following events: Disease progression (before surgery) as determined by the investigator with use of RECIST V1.1. Disease recurrence (local, regional, or distant) after surgery. Contralateral breast cancer. Second primary tumor. Death from any cause.
Overall survival (OS) | Time Frame: From Baseline to OS event or date last known to be alive (up to 10 years)
  OS was defined as the time from diagnosis to death from any cause.

OTHER OUTCOMES:
Percentage of Participants With At Least One Adverse Event During Treatment Period | From randomization to 30 days after completion of study treatment
  The percentage of participants who experienced at least one adverse event during study treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Abramson VG, Lehmann BD, Ballinger TJ, Pietenpol JA. Subtyping of triple-negative breast cancer: implications for therapy. Cancer. 2015 Jan 1;121(1):8-16. doi: 10.1002/cncr.28914. Epub 2014 Jul 16. PMID 25043972
- [Background] Cleator S, Heller W, Coombes RC. Triple-negative breast cancer: therapeutic options. Lancet Oncol. 2007 Mar;8(3):235-44. doi: 10.1016/S1470-2045(07)70074-8. PMID 17329194
- [Background] Scott LC, Mobley LR, Kuo TM, Il'yasova D. Update on triple-negative breast cancer disparities for the United States: A population-based study from the United States Cancer Statistics database, 2010 through 2014. Cancer. 2019 Oct 1;125(19):3412-3417. doi: 10.1002/cncr.32207. Epub 2019 Jul 8. PMID 31282032
- [Background] Bianchini G, Balko JM, Mayer IA, Sanders ME, Gianni L. Triple-negative breast cancer: challenges and opportunities of a heterogeneous disease. Nat Rev Clin Oncol. 2016 Nov;13(11):674-690. doi: 10.1038/nrclinonc.2016.66. Epub 2016 May 17. PMID 27184417
- [Background] Schott AF, Hayes DF. Defining the benefits of neoadjuvant chemotherapy for breast cancer. J Clin Oncol. 2012 May 20;30(15):1747-9. doi: 10.1200/JCO.2011.41.3161. Epub 2012 Apr 16. No abstract available. PMID 22508810
- [Background] Biswas T, Efird JT, Prasad S, Jindal C, Walker PR. The survival benefit of neoadjuvant chemotherapy and pCR among patients with advanced stage triple negative breast cancer. Oncotarget. 2017 Nov 20;8(68):112712-112719. doi: 10.18632/oncotarget.22521. eCollection 2017 Dec 22. PMID 29348858
- [Background] Chen VE, Gillespie EF, Zakeri K, Murphy JD, Yashar CM, Lu S, Einck JP. Pathologic response after neoadjuvant chemotherapy predicts locoregional control in patients with triple negative breast cancer. Adv Radiat Oncol. 2017 Feb 7;2(2):105-109. doi: 10.1016/j.adro.2017.01.012. eCollection 2017 Apr-Jun. PMID 28740920
- [Background] Gamucci T, Pizzuti L, Sperduti I, Mentuccia L, Vaccaro A, Moscetti L, Marchetti P, Carbognin L, Michelotti A, Iezzi L, Cassano A, Grassadonia A, Astone A, Botticelli A, Magnolfi E, Di Lauro L, Sergi D, Fuso P, Tinari N, Barba M, Maugeri-Sacca M, Landucci E, Conti F, Sanguineti G, De Tursi M, Iafrate G, Giordano A, Ciliberto G, Natoli C, Vici P. Neoadjuvant chemotherapy in triple-negative breast cancer: A multicentric retrospective observational study in real-life setting. J Cell Physiol. 2018 Mar;233(3):2313-2323. doi: 10.1002/jcp.26103. Epub 2017 Sep 27. PMID 28710865
- [Background] Loibl S, O'Shaughnessy J, Untch M, Sikov WM, Rugo HS, McKee MD, Huober J, Golshan M, von Minckwitz G, Maag D, Sullivan D, Wolmark N, McIntyre K, Ponce Lorenzo JJ, Metzger Filho O, Rastogi P, Symmans WF, Liu X, Geyer CE Jr. Addition of the PARP inhibitor veliparib plus carboplatin or carboplatin alone to standard neoadjuvant chemotherapy in triple-negative breast cancer (BrighTNess): a randomised, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):497-509. doi: 10.1016/S1470-2045(18)30111-6. Epub 2018 Feb 28. PMID 29501363
- [Background] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Background] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Background] Sharma P, Kimler BF, O'Dea A, Nye L, Wang YY, Yoder R, Staley JM, Prochaska L, Wagner J, Amin AL, Larson K, Balanoff C, Elia M, Crane G, Madhusudhana S, Hoffmann M, Sheehan M, Rodriguez R, Finke K, Shah R, Satelli D, Shrestha A, Beck L, McKittrick R, Pluenneke R, Raja V, Beeki V, Corum L, Heldstab J, LaFaver S, Prager M, Phadnis M, Mudaranthakam DP, Jensen RA, Godwin AK, Salgado R, Mehta K, Khan Q. Randomized Phase II Trial of Anthracycline-free and Anthracycline-containing Neoadjuvant Carboplatin Chemotherapy Regimens in Stage I-III Triple-negative Breast Cancer (NeoSTOP). Clin Cancer Res. 2021 Feb 15;27(4):975-982. doi: 10.1158/1078-0432.CCR-20-3646. Epub 2020 Nov 18. PMID 33208340
- [Background] Zhang L, Wu ZY, Li J, Lin Y, Liu Z, Cao Y, Zhang G, Gao HF, Yang M, Yang CQ, Zhu T, Cheng MY, Ji F, Li J, Wang K. Neoadjuvant docetaxel plus carboplatin vs epirubicin plus cyclophosphamide followed by docetaxel in triple-negative, early-stage breast cancer (NeoCART): Results from a multicenter, randomized controlled, open-label phase II trial. Int J Cancer. 2022 Feb 15;150(4):654-662. doi: 10.1002/ijc.33830. Epub 2021 Oct 7. PMID 34591977
- [Background] Chen XS, Nie XQ, Chen CM, Wu JY, Wu J, Lu JS, Shao ZM, Shen ZZ, Shen KW. Weekly paclitaxel plus carboplatin is an effective nonanthracycline-containing regimen as neoadjuvant chemotherapy for breast cancer. Ann Oncol. 2010 May;21(5):961-7. doi: 10.1093/annonc/mdq041. Epub 2010 Mar 8. PMID 20211870
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Buque A, Bloy N, Aranda F, Castoldi F, Eggermont A, Cremer I, Fridman WH, Fucikova J, Galon J, Marabelle A, Spisek R, Tartour E, Zitvogel L, Kroemer G, Galluzzi L. Trial Watch: Immunomodulatory monoclonal antibodies for oncological indications. Oncoimmunology. 2015 Mar 2;4(4):e1008814. doi: 10.1080/2162402X.2015.1008814. eCollection 2015 Apr. PMID 26137403
- [Background] Syn NL, Teng MWL, Mok TSK, Soo RA. De-novo and acquired resistance to immune checkpoint targeting. Lancet Oncol. 2017 Dec;18(12):e731-e741. doi: 10.1016/S1470-2045(17)30607-1. PMID 29208439
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Gaynor N, Crown J, Collins DM. Immune checkpoint inhibitors: Key trials and an emerging role in breast cancer. Semin Cancer Biol. 2022 Feb;79:44-57. doi: 10.1016/j.semcancer.2020.06.016. Epub 2020 Jul 2. PMID 32623044
- [Background] Makhoul I, Atiq M, Alwbari A, Kieber-Emmons T. Breast Cancer Immunotherapy: An Update. Breast Cancer (Auckl). 2018 May 30;12:1178223418774802. doi: 10.1177/1178223418774802. eCollection 2018. PMID 29899661
- [Background] Disis ML, Stanton SE. Triple-negative breast cancer: immune modulation as the new treatment paradigm. Am Soc Clin Oncol Educ Book. 2015:e25-30. doi: 10.14694/EdBook_AM.2015.35.e25. PMID 25993181
- [Background] Mittendorf EA, Philips AV, Meric-Bernstam F, Qiao N, Wu Y, Harrington S, Su X, Wang Y, Gonzalez-Angulo AM, Akcakanat A, Chawla A, Curran M, Hwu P, Sharma P, Litton JK, Molldrem JJ, Alatrash G. PD-L1 expression in triple-negative breast cancer. Cancer Immunol Res. 2014 Apr;2(4):361-70. doi: 10.1158/2326-6066.CIR-13-0127. Epub 2014 Jan 10. PMID 24764583
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] Schmid P, Cortes J, Dent R, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Untch M, Fasching PA, Cardoso F, Andersen J, Patt D, Danso M, Ferreira M, Mouret-Reynier MA, Im SA, Ahn JH, Gion M, Baron-Hay S, Boileau JF, Ding Y, Tryfonidis K, Aktan G, Karantza V, O'Shaughnessy J; KEYNOTE-522 Investigators. Event-free Survival with Pembrolizumab in Early Triple-Negative Breast Cancer. N Engl J Med. 2022 Feb 10;386(6):556-567. doi: 10.1056/NEJMoa2112651. PMID 35139274
- [Background] Mittendorf EA, Zhang H, Barrios CH, Saji S, Jung KH, Hegg R, Koehler A, Sohn J, Iwata H, Telli ML, Ferrario C, Punie K, Penault-Llorca F, Patel S, Duc AN, Liste-Hermoso M, Maiya V, Molinero L, Chui SY, Harbeck N. Neoadjuvant atezolizumab in combination with sequential nab-paclitaxel and anthracycline-based chemotherapy versus placebo and chemotherapy in patients with early-stage triple-negative breast cancer (IMpassion031): a randomised, double-blind, phase 3 trial. Lancet. 2020 Oct 10;396(10257):1090-1100. doi: 10.1016/S0140-6736(20)31953-X. Epub 2020 Sep 20. PMID 32966830
- [Background] Gianni L, Huang CS, Egle D, Bermejo B, Zamagni C, Thill M, Anton A, Zambelli S, Bianchini G, Russo S, Ciruelos EM, Greil R, Semiglazov V, Colleoni M, Kelly C, Mariani G, Del Mastro L, Maffeis I, Valagussa P, Viale G. Pathologic complete response (pCR) to neoadjuvant treatment with or without atezolizumab in triple-negative, early high-risk and locally advanced breast cancer: NeoTRIP Michelangelo randomized study. Ann Oncol. 2022 May;33(5):534-543. doi: 10.1016/j.annonc.2022.02.004. Epub 2022 Feb 17. PMID 35182721
- [Background] Loibl S, Untch M, Burchardi N, Huober J, Sinn BV, Blohmer JU, Grischke EM, Furlanetto J, Tesch H, Hanusch C, Engels K, Rezai M, Jackisch C, Schmitt WD, von Minckwitz G, Thomalla J, Kummel S, Rautenberg B, Fasching PA, Weber K, Rhiem K, Denkert C, Schneeweiss A. A randomised phase II study investigating durvalumab in addition to an anthracycline taxane-based neoadjuvant therapy in early triple-negative breast cancer: clinical results and biomarker analysis of GeparNuevo study. Ann Oncol. 2019 Aug 1;30(8):1279-1288. doi: 10.1093/annonc/mdz158. PMID 31095287